CLINICAL TRIAL: NCT03349034
Title: Role of Continuous Local Infusion of Ropivacaine for Post-Operative Pain Management in Patients Receiving Osseocutaneous Free Flaps
Brief Title: Local Infusion of Ropivacaine for Post-Op Pain Control After Osseocutaneous Free Flaps
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Brett Miles, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: GCO 17-1391
Record Dates: First submitted 2017-11-17; First posted 2017-11-21 (Actual); Results first posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-10

CONDITIONS: Head and Neck Cancer; Free Tissue Transfer
Keywords: Local anesthetics; Randomized Control Trial; Free tissue transfer; Head and neck; Microvascular; Postoperative Pain
MeSH Terms: conditions — Head and Neck Neoplasms; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: The study is a double-blind prospective randomized placebo controlled trial wherein patients undergoing osseocutaneous free flap surgery are randomized to receive continuous infusion of Ropivacaine or normal saline (placebo) via local infusion catheter, which will be placed intraoperatively at the time of donor site closure. Outcomes are tracked and assessed for the first 48 hours post-operatively - median post-operative pain assessed via VAS every 8 hours, total analgesic used (all patients receive Tylenol 650 and dilaudid PCA post-operatively), physical therapy outcomes assessed on post-operative day two, and a patient satisfaction survey.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Local Ropivicaine Infusion
  Interventions: Drug: Ropivicaine
- Control Group (Placebo Comparator): Local Saline Infusion
  Interventions: Drug: Local Saline Infusion

INTERVENTIONS:
Drug: Ropivicaine — Patients will be randomized to receive a local continuous infusion of 6 ml/hr of 0.2% Ropivacaine via On-Q infusion pump, at the donor site, for the first 48 hours of the postoperative period.
  Arms: Test Group
Drug: Local Saline Infusion — Patients will be randomized to receive a local continuous infusion of 6 ml/hr of 0.9% normal saline via On-Q infusion pump, at the donor site, for the first 48 hours of the postoperative period.
  Arms: Control Group

SUMMARY:
Head and neck oncologic surgery often requires the use of free tissue transfer, or microvascular reconstruction, to reconstruct defects created by tumor resections. Although there are several techniques for the reconstruction of defects, resection of large tumors leave defects that require the transfer of vascularized tissue from one part of the body to repair the defect. For example, the removal of a segment of diseased mandible requires free tissue transfer containing the component parts - skin, muscle, and bone - to reconstruct the deficit created by the resection of the tumor. Over the years, microvascular surgeons have focused their attention on maximizing the success of these technically difficult surgeries. However, now, with free flap reconstruction rates in excess of 95%, surgeons are afforded the opportunity to turn their focus toward the morbidities associated with these surgeries. While much has been published about donor site wound healing, pain control in the post-operative period has largely been neglected in the head and neck reconstruction literature. Systemic analgesia with opioids is standard of care, which has been shown to lead to increased confusion, significantly increased length of stay and increased risk of pulmonary complications. In addition, it has been shown that early mobilization and optimal wound care can decrease donor site morbidity.

In this study the clinical team aims to better control donor site pain utilizing local, targeted analgesia to relieve pain at the donor site for osseocutaneous free-flaps. To reduce confounding and bias, the study will be a double-blind prospective randomized placebo controlled trial wherein patients undergoing osseocutaneous free flap surgery will be randomized to receive continuous infusion of ropivacaine or normal saline (placebo) via local continuous infusion catheter, which will be placed intraoperatively at the time of donor site closure. Patients' pain will be monitored for the first 48hrs after surgery. Donor site and global pain at rest will be evaluated every 8 hours for the first two postoperative days using a visual analogue pain scale (VAS). Essentially, there is a 100 millimeter line drawn on a piece of paper, with "no pain" marking the left end of the line and "worst pain" marking the right end of the line. Subjects mark with a pen along the line where pain is felt fits along that continuum. A researcher then measures how far along the line that mark is placed and then it is recorded. Median daily opiate use via PCA will also be tracked. Donor site-specific range of motion and strength will be assessed with a formal physical therapy evaluation on post-operative day 2 or soonest non-holiday weekday. Information on patient satisfaction, time to ambulation, and length of stay will also be collected. Subgroup analysis will be performed.

DETAILED DESCRIPTION:
Procedures involved in this study include:

- Intraoperatively, following procurement of the fibula or scapula bone graft and at the time of surgical wound closure, all patients will receive the placement of a continuous infusion catheter into the donor site wound bed. The infusion reservoir will be connected to a catheter-based On-Q pump, and the catheter will be placed in the donor site. A stab incision separate from the surgical wound will be used to bring the catheter through the skin. Patients will be randomized to receive 6 ml/hr of 0.2% Ropivacaine or 6 ml/hr of normal saline via the infusion reservoir. The catheter will be left in place with continuous infusion for first 48 hours of the post-operative period. The catheters will be removed by the housestaff on POD2. There is minimal risk to removing the OnQ catheter. Any opening in the skin will be covered with gauze to allow primary healing. Solutions of saline and ropivacaine will be prepared and made available for infusion by the Mount Sinai Pharmacy. Solutions will be blinded, and identical in appearance. Patients will be assigned to ropivacaine or saline intervention by the research pharmacy through coded envelopes. Patients, physicians, nurses, and research personnel will be blinded to treatment assignment. Every 8 hours for the first 48 hours, patients will be asked to complete a visual analogue scale (VAS) for reporting their pain. The VAS will be performed six times over the course of the 48hrs. These will be performed during regular flap check monitoring, to ensure patients are not disrupted additional times throughout the day for this study. Patients will otherwise receive standard of care pain management, including Tylenol 650 q6hr standing as well as a dilaudid PCA set to low-dose, opioid naïve. On post-operative day 2 patient will receive a physical therapy evaluation.

Prior to discharge from the hospital, the study subjects will be asked to complete a brief survey (APS-POQ-R Pain Survey) regarding their experience, with regard to pain management.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving osseocutaneous free tissue transfer regardless of the indication for free tissue transfer.

This includes osseocutaneous tissue from fibula and scapula

* Age ≥ 18

Exclusion Criteria:

* Patients unable to understand the research protocol and/or provide informed consent
* Patients under the age of 18
* Patients with a history of allergic reaction to Ropivacaine or other local amide anesthetics
* Patients whose participation in this trial would require exclusion from participation in another clinical research trial related to the patient's malignant diagnosis.
* Patients with previous pain disorders or drug abuse requiring chronic narcotic use.
* Vulnerable populations (adults unable to consent, individuals who are not yet adults, wards of the state, prisoners)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Genden, MD, Study Chair — Icahn School of Medicine at Mount Sinai; Brett Miles, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blumenthal S, Dullenkopf A, Rentsch K, Borgeat A. Continuous infusion of ropivacaine for pain relief after iliac crest bone grafting for shoulder surgery. Anesthesiology. 2005 Feb;102(2):392-7. doi: 10.1097/00000542-200502000-00023. PMID 15681956
- [Background] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233
- [Background] Oderda GM, Said Q, Evans RS, Stoddard GJ, Lloyd J, Jackson K, Rublee D, Samore MH. Opioid-related adverse drug events in surgical hospitalizations: impact on costs and length of stay. Ann Pharmacother. 2007 Mar;41(3):400-6. doi: 10.1345/aph.1H386. Epub 2007 Mar 6. PMID 17341537
- [Background] Singh K, Samartzis D, Strom J, Manning D, Campbell-Hupp M, Wetzel FT, Gupta P, Phillips FM. A prospective, randomized, double-blind study evaluating the efficacy of postoperative continuous local anesthetic infusion at the iliac crest bone graft site after spinal arthrodesis. Spine (Phila Pa 1976). 2005 Nov 15;30(22):2477-83. doi: 10.1097/01.brs.0000186323.11285.b1. PMID 16284583
- [Derived] Roof S, Ferrandino R, Eden C, Khelemsky Y, Teng M, Genden E, DeMaria S Jr, Miles BA. Local infusion of ropivacaine for pain control after osseous free flaps: Randomized controlled trial. Head Neck. 2021 Apr;43(4):1063-1072. doi: 10.1002/hed.26562. Epub 2021 Feb 23. PMID 33619855

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants undergoing osseocutaneous fibula or scapular tip free flaps for head and neck reconstructionwere enrolled from September 2017 and September 2019.
Groups:
- Saline Placebo: Local Saline Infusion: Patients randomized to receive a local continuous infusion of 6 ml/hr of 0.9% normal saline via On-Q infusion pump, at the donor site, for the first 48 hours of the postoperative period.
- Ropivacaine: Local Ropivicaine Infusion: Patients randomized to receive a local continuous infusion of 6 ml/hr of 0.2% Ropivacaine via On-Q infusion pump, at the donor site, for the first 48 hours of the postoperative period.
Period: Overall Study
Arm/Group | Saline Placebo | Ropivacaine
Started | 12 | 12
Completed | 8 | 10
Not Completed | 4 | 2
Not completed — catheters dislodged during transport | 2 | 0
Not completed — intubated for >48 hrs following surgery | 1 | 1
Not completed — soft tissue flap used | 1 | 0
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline Placebo | Ropivacaine | Total
Number analyzed (Participants) | 8 | 10 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (11.6) | 67.1 (13.7) | 66.2 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 8 | 8 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.2 (4.81) | 28.7 (4.39) | 28.0 (4.51)
ASA Physical Status Classification System [Mean (Standard Deviation); unit: units on a scale] — American Society of Anesthesiologists Physical Status Classification I - A normal healthy patient II - A patient with mild systemic disease III - A patient with severe systemic disease IV - A patient with severe systemic disease that is a constant threat to life V - A moribund patient who is not expected to survive without the operation VI - A declared brain-dead patient whose organs are being removed for donor purposes
  units on a scale | 2.88 (0.35) | 3.10 (0.32) | 3.0 (0.34)
Pack Years [Mean (Standard Deviation); unit: cigarettes per day for 1 year] — calculated by multiplying the number of packs of cigarettes smoked per day by the number of years the person has smoked.
  cigarettes per day for 1 year | 7.75 (15.1) | 7.30 (10.1) | 7.5 (12.2)
Smoking at Diagnosis [Count of Participants; unit: Participants] | 0 | 1 | 1
Number of participants with Alcohol Abuse [Count of Participants; unit: Participants] | 1 | 0 | 1
Number of participants with Diabetes Mellitus [Count of Participants; unit: Participants] | 3 | 4 | 7
Tumor Type [Count of Participants; unit: Participants]
  squamous cell carcinoma (SCC) | 4 | 6 | 10
  Benign | 4 | 4 | 8
Primary Site/Procedure [Count of Participants; unit: Participants]
  Maxilla/Maxillectomy | 5 | 2 | 7
  Mandible/Mandibulectomy | 3 | 8 | 11
Flap Type [Count of Participants; unit: Participants]
  Scapula | 4 | 6 | 10
  Fibula | 4 | 4 | 8
Previous Treatment [Count of Participants; unit: Participants]
  History of Radiation Therapy | 1 | 3 | 4
  History of Chemotherapy | 1 | 2 | 3
Length of Stay [Mean (Standard Deviation); unit: days] | 11.5 (3.89) | 13.8 (6.34) | 12.8 (5.37)

OUTCOME MEASURES:

1. Primary Outcome: Post-Operative Pain at Donor-Site
Description: Pain assessed every 8 hours for the first 48 hours using a visual analogue pain scale at rest. A visual analogue pain scale is a validated pain measure. Essentially, there is a 100 millimeter line drawn on a piece of paper, with "no pain" marking the left end of the line and "worst pain" marking the right end of the line. Subjects mark with a pen along the line where pain is felt fits along that continuum. A researcher then measures how far along the line that mark is placed and then it is recorded. Full scale from 0-100, higher score indicates more pain.
Time Frame: 8, 16, 24, 32, 40 and 48 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Saline Placebo | Ropivacaine
Number analyzed (Participants) | 8 | 10
score on a scale
  8 hour | 52.40 (25.33) | 41.14 (28.30)
  16 hour | 41.00 (33.20) | 40.88 (31.46)
  24 hour | 23.33 (29.28) | 45.67 (24.87)
  32 hour | 25.67 (27.28) | 37.44 (31.11)
  40 hour | 30.12 (22.29) | 42.11 (30.64)
  48 hour | 28.75 (21.72) | 30.60 (28.30)

2. Primary Outcome: Post-Operative Pain - Global Pain
Description: as for outcome 1
Time Frame: 8, 16, 24, 32, 40 and 48 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Saline Placebo | Ropivacaine
Number analyzed (Participants) | 8 | 10
score on a scale
  8 hour | 44.00 (28.55) | 40.14 (32.25)
  16 hour | 27.50 (23.18) | 26.56 (27.03)
  24 hour | 31.83 (21.25) | 41.56 (30.33)
  32 hour | 24.17 (25.91) | 35.67 (32.39)
  40 hour | 21.88 (20.36) | 33.60 (28.76)
  48 hour | 20.38 (13.43) | 37.40 (35.50)

3. Secondary Outcome: Opioid Consumption
Description: All subjects receive standing tylenol 650mg every 6 hours as well as a dilaudid PCA set for low-dose, opioid-naive patients for the first 48 hours post-operatively. Total opioid consumption for each subject during the first 48 hours is recorded measured in oral morphine equivalents (OME).
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: OME
Arm/Group | Saline Placebo | Ropivacaine
Number analyzed (Participants) | 8 | 10
OME | 119.75 (145.92) | 91.20 (132.14)

4. Secondary Outcome: Range of Motion
Description: At 48 hours all subjects will receive a physical therapy evaluation. Range of motion will be measured in degrees
Time Frame: 48 hours
Population: Data not collected
Groups:
- Saline Placebo: Local Saline Infusion: Patients will be randomized to receive a local continuous infusion of 6 ml/hr of 0.9% normal saline via On-Q infusion pump, at the donor site, for the first 48 hours of the postoperative period.
- Ropivacaine: Local Ropivicaine Infusion: Patients will be randomized to receive a local continuous infusion of 6 ml/hr of 0.2% Ropivacaine via On-Q infusion pump, at the donor site, for the first 48 hours of the postoperative period.
Arm/Group | Saline Placebo | Ropivacaine
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Distance Ambulated
Description: At 48 hours all subjects received a physical therapy evaluation. Distance ambulated measured in feet.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Saline Placebo | Ropivacaine
Number analyzed (Participants) | 8 | 10
feet | 152 (111.9) | 80 (67.08)

6. Secondary Outcome: Strength
Description: At 48 hours all subjects received a physical therapy evaluation. Strength measured on a standard neurological 5 point scale: 0 = Complete Paralysis to 5 = Normal Power.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Saline Placebo | Ropivacaine
Number analyzed (Participants) | 8 | 10
score on a scale | 2.67 (0.82) | 2.20 (1.10)

7. Secondary Outcome: American Pain Society-Patient Outcome Questionnaire - (APS-POQ-R)
Description: Pain question on APS-POQ-R - A standardized pain satisfaction survey distributed to subjects at 48 hours rating their overall satisfaction with postoperative pain management. a 16-item questions measured on a 10-point numeric likert scale, with higher scores indicating more pain. Total range from 0 (no pain) to 200 (severe pain).
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Saline Placebo | Ropivacaine
Number analyzed (Participants) | 8 | 10
score on a scale | 6.0 (2.39) | 4.3 (1.34)

ADVERSE EVENTS:
Time Frame: 48 hours post surgery
Arm/Group | Saline Placebo | Ropivacaine
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 0/8 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-19): https://cdn.clinicaltrials.gov/large-docs/34/NCT03349034/Prot_SAP_000.pdf